CLINICAL TRIAL: NCT00302614
Title: The Role of Clinical Parameters in Predicting the Severity of Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461701256
Record Dates: First submitted 2006-03-12; First posted 2006-03-14 (Estimated); Last update posted 2006-03-14 (Estimated); Status verified 2005-12

CONDITIONS: Obstructive Sleep Apnea; Snoring
Keywords: obstructive sleep apnea; snoring; collapsibility; upper airway
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Retrospective

SUMMARY:
Investigate the role of clinical parameters in predicting the severity of obstructive sleep apnea

DETAILED DESCRIPTION:
During the last two decades the obstructive sleep apnea syndrome (OSAS) has been increasingly recognized as a distinct clinical entity. This condition is caused by recurrent upper airway obstruction during sleep, is manifest as loud snoring, arterial oxygen desaturation, sleep fragmentation, and excessive daytime sleepiness1,2. Epidemiological series have shown that about 4% of the population suffers from symptomatic OSAS that requires treatment3-5. OSAS is associated with increased rates of many chronic diseases6,7 and is a serious and potentially life-threatening disorder that is far more common than generally believed. Thus, untreated OSAS may pose a significant public health problem8. Epidemiological data demonstrating the relationship between OSAS and cardiovascular morbidity highlight the potential importance of early recognition and treatment9.

The mechanisms responsible for upper airway obstruction in patients with OSAS are highly complicated and as yet not fully understood. Several causes for OSAS have been suggested. It appears to result from a variable combination of anatomic and pathophysiologic factors, some of which may be under genetic control10. The relaxation of upper airway musculature has been studied in relation to OSAS11-13. Anatomic narrowing of the upper airway as a result of alterations in craniofacial morphology or soft tissue enlargement, the Bernoulli effect, sleep posture, age, male gender, and adipose tissue in the pharynx have been suggested in the etiology of OSAS14-17.

Several studies have suggested that ethnicity may be an important risk factor in OSAS17-20. Recent reports have suggested that Asian subjects with OSAS have a greater severity of illness compared with white subjects21,22. Some studies reported that obesity is the strongest risk factor for OSAS in middle-aged adults3,23,24. However, we have treated many non-obese Taiwanese young adults with severe OSAS. Previous researches have suggested that there may be differences in obesity and craniofacial anatomy as risk factors between Asians and whites25 and that the etiology of OSAS in obese patients may be different from that in non-obese patients16,26,27. It is still unclear whether there are differences in clinical evaluation parameters between non-obese Asian patients with severe OSAS and simple snoring.

We hypothesized that there are predictor factors in routine clinical examinations for diagnosis of OSAS in non-obese young adult patients. Therefore, the objectives of this study are to compare the clinical parameters in non-obese patients with severe OSAS with those of simple snorers and to find the risk factors for OSAS in a non-obese young adult Taiwanese population.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnea or snoring patients

Exclusion Criteria:

* Patients with any concurrent medical illnesses except hypertension

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100
Dates: Start 2006-01; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Ting Tan, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan